CLINICAL TRIAL: NCT06196112
Title: Localization of Vasculonervous Structures in Tibial Nerve Neuromodulation: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Irene Lázaro Navas, Physiotherapy, PhD, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Other Study IDs: 115/23
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Tibial Nerve; Healthy Volunteers
Keywords: tibial arteries; ultrasonography; Pelvic Floor Disorders; Transcutaneous Electric Nerve Stimulation
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tibial nerve neuromodulation is an effective and widely used technique in various pelvic floor dysfunctions. There are two approaches described in scientific literature to perform this technique: transcutaneous and percutaneous. However, there is no consensus on the execution of these techniques, as the location of the tibial nerve in relation to other anatomical structures like the tibia has not been described. The findings of this research could serve as a basis for the implementation and development of protocols aimed at improving the technique of posterior tibial neuromodulation.

DETAILED DESCRIPTION:
Design: A cross-sectional observational study at the Physiotherapy Unit of the Ramón y Cajal University Hospital.

The main objective of this study is to determine the location and size of tibial vasculonervous structures (nerve, artery, and vein) in relation to the tibia and skin using ultrasound in healthy subjects Methods: Healthy subjects will participate, and sociodemographic data (age, sex, weight, height) will be collected. Subsequently, various measurements of the right tibial vasculonervous structures will be obtained through ultrasound A single examiner with over 5 years of experience in ultrasound will perform the measurements.

Significance of the research: Knowledge of the position and size of the tibial vasculonervous bundle could be useful to justify and standardize transcutaneous and percutaneous approaches in tibial nerve neuromodulation. This would improve the safety of the technique, avoiding adverse events resulting from the intervention

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects over 18 years of age

Exclusion Criteria:

* Previous fracture of the distal end of the right tibia
* Previous vascular pathology of the distal end of the right tibia
* Previous nervous condition of the distal end of the right tibia
* Previous surgical intervention of the distal end of the right tibia
* Ongoing oncological process of the distal end of the right tibia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing treatment at the Rehabilitation Service and among the workers of Ramón y Cajal University Hospital who meet the selection criteria
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Tibial Distance (TD) to the tibial nerve | Day 1
  Subjects will be placed in a right lateral decubitus position on a bed. Seven marks will be made with a dermal marker from the lower edge of the right tibial malleolus, following the medial edge of the tibial bone in the cranial direction. Measurements will be taken at 2, 4, 5, 6, 8, 10, and 12 cm with respect to the lower edge of the tibial malleolus. The most superficial aspect of the tibia will be considered for the measurements.
  The measurements will be performed using an ultrasound machine (ALPINIONⓒ, Seoul, South Korea, model ECUBE 8LEⓇ) with a linear probe L3-12T (frequency range 3-12 MHz), using the Rehabilitative Ultrasound Imaging (RUSI) method.
  The distance will be measured using a caliper by drawing a straight line from the most medial aspect of the tibia to the most anterior aspect of the nerve, taking into consideration the outer edge of the tibial nerve wall. This will be analyzed at each of the 7 marks previously described
Tibial Distance (TD) to the tibial artery | Day 1
  Subjects will be placed in a right lateral decubitus position on a bed. Seven marks will be made with a dermal marker from the lower edge of the right tibial malleolus, following the medial edge of the tibial bone in the cranial direction. Measurements will be taken at 2, 4, 5, 6, 8, 10, and 12 cm with respect to the lower edge of the tibial malleolus. The most superficial aspect of the tibia will be considered for the measurements.
  The measurements will be performed using an ultrasound machine (ALPINIONⓒ, Seoul, South Korea, model ECUBE 8LEⓇ) with a linear probe L3-12T (frequency range 3-12 MHz), using the Rehabilitative Ultrasound Imaging (RUSI) method.
  The distance will be measured using a caliper by drawing a straight line from the most medial aspect of the tibia to the most anterior aspect of the artery, taking into consideration the outer edge of the tibial artery wall. This will be analyzed at each of the 7 marks previously described
Tibial Distance (TD) to the tibial vein | Day 1
  Subjects will be placed in a right lateral decubitus position on a bed. Seven marks will be made with a dermal marker from the lower edge of the right tibial malleolus, following the medial edge of the tibial bone in the cranial direction. Measurements will be taken at 2, 4, 5, 6, 8, 10, and 12 cm with respect to the lower edge of the tibial malleolus. The most superficial aspect of the tibia will be considered for the measurements.
  The measurements will be performed using an ultrasound machine (ALPINIONⓒ, Seoul, South Korea, model ECUBE 8LEⓇ) with a linear probe L3-12T (frequency range 3-12 MHz), using the Rehabilitative Ultrasound Imaging (RUSI) method.
  The distance will be measured using a caliper by drawing a straight line from the most medial aspect of the tibia to the most anterior aspect of the vein, taking into consideration the outer edge of the tibial vein wall. This will be analyzed at each of the 7 marks previously described

SECONDARY OUTCOMES:
Horizontal Tibial Distance to the tibial nerve | Day 1
  The horizontal distance will be collected by drawing a perpendicular line with the caliper from the most medial aspect of the tibia to the most anterior aspect of the nerve, taking into consideration the outer edge of the tibial nerve wall. The measurement will be taken at each of the 7 marks previously described. This measurement will allow for an extrapolation in the implementation of percutaneous techniques
Horizontal Tibial Distance to the tibial artery | Day 1
  The horizontal distance will be collected by drawing a perpendicular line with the caliper from the most medial aspect of the tibia to the most anterior aspect of the artery tibial, taking into consideration the outer edge of the tibial artery wall. The measurement will be taken at each of the 7 marks previously described. This measurement will allow for an extrapolation in the implementation of percutaneous techniques
Horizontal Tibial Distance to the tibial vein | Day 1
  The horizontal distance will be collected by drawing a perpendicular line with the caliper from the most medial aspect of the tibia to the most anterior aspect of the vein, taking into consideration the outer edge of the tibial vein wall. The measurement will be taken at each of the 7 marks previously described. This measurement will allow for an extrapolation in the implementation of percutaneous techniques
Depth of the tibial nerve | Day 1
  Using the ultrasound machine and considering a caliper perpendicular from the most superficial aspect of the skin to the most superficial aspect of the epineurium at each of the 7 previously described marks
Cross-sectional area of the tibial nerve | Day 1
  The cross-sectional area of the nerve will be measured at each of the 7 marks described above using the ultrasound
Cross-sectional area of the tibial artery | Day 1
  The cross-sectional area of the artery will be measured at each of the 7 marks described above using the ultrasound
Cross-sectional area of the tibial vein | Day 1
  The cross-sectional area of the vein will be measured at each of the 7 marks described above using the ultrasound
Overlap between each structure | Day 1
  The overlap between the tibial nerve, artery, and vein will be described at each of the 7 marks previously mentioned
Variability of the tibial vessels | Day 1
  The number of arteries and veins present will be recorded at each of the 7 marks previously described

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

REFERENCES:
- [Derived] Lazaro-Navas I, Cervera-Cano M, Pecos-Martin D, Lopez-Gonzalez L, Valcarcel-Linares D. Ultrasound Evaluation of Tibial Vasculonervous Structures for Tibial Nerve Neuromodulation: A Cross-Sectional Study. Neuromodulation. 2025 Dec;28(8):1318-1326. doi: 10.1016/j.neurom.2025.07.010. Epub 2025 Sep 11. PMID 40932423